CLINICAL TRIAL: NCT01314937
Title: Improving Early Childhood Growth and Development in Resource-poor LMICs by Incorporating Deworming in Integrated Child Health Care
Brief Title: The Effect of a Deworming Intervention to Improve Early Childhood Growth and Development in Resource-poor Areas
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: McGill University (Other); Asociacion Civil Selva Amazonica (Other); World Health Organization (Other); Thrasher Research Fund (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Theresa Gyorkos, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-242-PED
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Malnutrition; Intestinal Diseases, Parasitic
Keywords: preschool-age children; soil-transmitted helminths; growth; development; deworming
MeSH Terms: conditions — Malnutrition; Intestinal Diseases, Parasitic | interventions — Mebendazole; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Deworming at 12 months of age (Experimental)
  Interventions: Drug: Mebendazole; Other: Usual care
- Deworming at 18 months of age (Experimental)
  Interventions: Drug: Mebendazole; Other: Usual care
- Deworming at 12 and 18 months of age (Experimental)
  Interventions: Drug: Mebendazole; Other: Usual care
- Usual care (Placebo Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Drug: Mebendazole — Single-dose 500 mg mebendazole tablet
  Other Names: Vermox, Nemasole, Pantelmin
  Arms: Deworming at 12 and 18 months of age; Deworming at 12 months of age; Deworming at 18 months of age
Other: Usual care — Routine child health interventions (e.g. age-specific immunizations, supplementations, etc.)
  Other Names: Standard of care, routine health care services

SUMMARY:
Worldwide, over 2 billion people suffer from worm infections in developing countries. These infections are especially damaging to the health of children, resulting in both short-term and lifelong disability. Older children with worm infections are more likely to be stunted, underweight, vulnerable to other illnesses and perform poorly in school compared to non-infected children. Large-scale deworming programs in school-age children are therefore recommended by the World Health Organization (WHO). WHO also recommends deworming of preschool-age children (as of 12 months of age) in these areas; however, the benefits of deworming, especially in the 12-24 month age group, have been inadequately studied. This knowledge is urgently needed as studies show that all children have a similar potential for healthy growth and development, provided that appropriate nutrition and health interventions are given in the critical window of opportunity before the age of two.

Therefore, the investigators are proposing to undertake a randomized controlled trial to determine the effect of deworming program for improving growth and development in children between 12 and 24 months of age. Our results will provide solid rigorous evidence on if, when, and how often, deworming should be integrated into routine child health care packages provided by Ministries of Health in the 130 countries in the world where worm infections are endemic.

DETAILED DESCRIPTION:
Worldwide, over 2 billion people suffer from worm infections (hookworm, Ascaris and Trichuris, collectively referred to as soil-transmitted helminths (STHs)) in developing countries. STHs contribute to the overwhelming burden of poverty and deprivation in areas where adverse health, social, economic, education and other related factors predominate. STH infection in childhood results in short-term and lifelong disability, including malnutrition (e.g. underweight, stunting and wasting), cognitive impairment and increased susceptibility to other infection, among others. Mass deworming programs in school-age children are recommended by the World Health Organization (WHO). WHO also recommends deworming of preschool children (as of 12 months of age) in endemic areas; however, the benefits of deworming on improving growth and development, especially in the 12-24 month age group, have been inadequately studied. This knowledge is crucial because, with appropriate nutrition and health interventions, all children have a similar potential for healthy growth and development, provided that such interventions occur in the critical window of opportunity before the age of two.

Therefore, this double-blind randomized controlled trial will assess the benefit of deworming (mebendazole), integrated into routine child health care visits in a highly STH-endemic area (Iquitos, Peru), on the primary outcome of weight gain. Timing, frequency and impact of deworming will be considered. A total of 1760 children will be recruited at their routine 12-month check-up visit and randomly assigned to one of four intervention groups: Group 1 will receive usual care and mebendazole (single dose 500 mg) at their 12-month visit and usual care and a placebo tablet at their 18-month visit; Group 2 will receive usual care and a placebo tablet at their 12-month visit and usual care and mebendazole at their 18-month visit; Group 3 will receive usual care and mebendazole at both their 12-month and 18-month visit; and Group 4 will receive usual care and placebo at both their 12-month and 18-month visit. Usual care will consist of age-appropriate immunizations, supplements and other Peruvian Ministry of Health-recommended interventions. All children will be followed up to their 24-month visit and all will be given mebendazole at that time.

Additional secondary outcomes include length gain, motor and cognitive development and STH prevalence and intensity.

Improving child health is a priority area in global health research and a focus of the Millennium Development Goals. Early preschool-age children are at the most critical stage of growth and development and have been neglected in deworming programs. It is anticipated that the results will inform evidence-based policy on the provision of an integrated health package for young children in endemic areas and ultimately contribute to the reduction of health inequities in this vulnerable group.

ELIGIBILITY:
Inclusion Criteria:

* children attending any one of the participating study health centres for their routine 12-month growth and development visit
* children living in or near the study area

Exclusion Criteria:

* children who are attending the clinic for suspected STH infection
* children who have received deworming treatment in the six months prior to randomization
* parents planning to move outside of the study area within the next 12 months
* children under 12 months of age or 14 months of age or older
* children with serious congenital or chronic medical conditions and who would be considered by the attending staff not to benefit from deworming

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1760 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Mean (± standard deviation) weight gain (kg) | from 12 to 24 months of age
  Weight will be measured at baseline (12 months of age), and follow-up (18 and 24 months of age) to assess the effect of the deworming intervention on growth (in terms of weight)

SECONDARY OUTCOMES:
Mean (± standard deviation) height gain (cm) | from 12 to 24 months of age
  Height will be measured at baseline (12 months of age) and at follow-up (18 and 24 months of age) to evaluate the effect of the deworming intervention on growth (in terms of height)
Mean (± standard deviation) of the cognitive test score | from 12 to 24 months of age
  Cognitive development will be assessed using the Bayley Scale of Infant Development. This scale provides a raw score and standardized score based on age-specific abilities. This will be measured at both baseline (12 months of age) and follow-up (at 24 months of age) to evaluate the effects of the deworming intervention on cognitive development.
Soil-transmitted helminth infection (Ascaris, Trichuris or hookworm) - prevalence (%) and intensity (mean eggs per gram) | from 12 to 24 months of age
  Soil-transmitted helminth (STH) infection will be assessed from stool samples provided by participants. The Kato-Katz technique will be used to provide both an estimate of prevalence of each STH (e.g. % positive for each Ascaris, Trichuris, and/or hookworm) as well as an estimate of intensity of each STH (measured as mean eggs per gram of stool). This will be measured at baseline (12 months of age) and follow-up (18 and 24 months of age) to evaluate the effect of the deworming intervention on parasite prevalence and intensity.
Mean (± standard deviation) of the motor test score | from 12 to 24 months of age
  Fine motor development will be assessed using the Bayley Scale of Infant Development. This scale provides a raw score and standardized score based on age-specific abilities. This will be measured at both baseline (12 months of age) and follow-up (at 24 months of age) to evaluate the effects of the deworming intervention on motor development.
Mean (± standard deviation) of the language test score | from 12 to 24 months of age
  Receptive and expressive language development will be assessed using the Bayley Scale of Infant Development. This scale provides a raw score and standardized score based on age-specific abilities. This will be measured at both baseline (12 months of age) and follow-up (at 24 months of age) to evaluate the effects of the deworming intervention on language development.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa W Gyorkos, PhD, Principal Investigator — McGill University; Martin Casapia, MD, MPH, Principal Investigator — Asociacion Civil Selva Amazonica
Locations (1):
- Asociacion Civil Selva Amazonica, Iquitos, Loreto, Peru

REFERENCES:
- [Derived] Joseph SA, Casapia M, Montresor A, Rahme E, Ward BJ, Marquis GS, Pezo L, Blouin B, Maheu-Giroux M, Gyorkos TW. The Effect of Deworming on Growth in One-Year-Old Children Living in a Soil-Transmitted Helminth-Endemic Area of Peru: A Randomized Controlled Trial. PLoS Negl Trop Dis. 2015 Oct 1;9(10):e0004020. doi: 10.1371/journal.pntd.0004020. eCollection 2015. PMID 26426270